CLINICAL TRIAL: NCT04825418
Title: Beneficial Effect of Therapeutic Hypothermia Plus Hemicraniectomy Compared With Hemicraniectomy Alone in Patients With Malignant Cerebral Infarction (BETHLeHAM Study) - Prospective, Open, Single-arm, Multicenter Phase II Study
Brief Title: Beneficial Effect of Hypothermia Plus Hemicraniectomy Compared With Hemicraniectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Bard Medical Division C.R. Bard Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BETHLeHAM
Record Dates: First submitted 2021-03-28; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-01

CONDITIONS: Hypothermia
Keywords: therapeutic hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapeutic Hypothermia Group (Experimental): Therapeutic hypothermia using surface cooling device (Arctic Sun) Decompressive Hemicraniectomy care based on international guidelines except therapeutic hypothermia using surface cooling device.
  Interventions: Device: Artic Sun

INTERVENTIONS:
Device: Artic Sun — 1. Induction phase A. Temperature using by esophageal or bladder thermometer. B. Application of a surface cooling device (Arctic Sun) C. Target temperature: 35 ± 0.5 °C D. Induction should be initiated as soon as possible after surgery (less than 6 hours)
  2. Maintain phase A. Maintain duration : at least 72 hours and duration can be prolonged according to patient's clinical status B. Use the bedside shivering assessment scale (BSAS) and anti-shivering protocol C. Neuromuscular blocker can be used according to the discretion of the attending physician D. Lung-protective ventilation strategies including low-tidal volume are recommended E. Prophylactic antibiotics can be used to prevent pneumonia during hypothermia
  3. Rewarming phase A. Rewarming rate: 0.05 - 0.1 ℃/hr (about 20 - 40 hours) to 37 ℃
  Other Names: Therapeutic Hypothermia Group

SUMMARY:
To study safety and feasibility of mild therapeutic hypothermia after decompressive hemicraniectomy compared with hemicraniectomy alone in patients with malignant cerebral infarction

DETAILED DESCRIPTION:
The current clinical trial is an investigator-initiated one, and it is conducted under the multi-center, single arm, open-label, prospective design. The subject meeting inclusion/exclusion criteria will be assigned to treatment group.

The subjects of treatment group should be initiated hypothermia therapy as soon as possible after surgery (less than 6 hours). It can be duration at least 72 hours according to subject status. Also process of recovery temperature period will be allowed within 20-40 hours. After 6 month, 12 month of the onset of symptom, mRS score are measured. This is followed by closure of clinical trial.

ELIGIBILITY:
Inclusion Criteria:

A. Written informed consent obtained from the patient or his/her legally acceptable representative B. Acute ischemic stroke within middle cerebral artery or internal carotid artery occlusion

* Regardless of anterior cerebral artery (ACA) or posterior cerebral artery (PCA) involvement C. Patients of both sexes aged ≥ 19 years and ≤ 82 years D. NIHSS score ≥ 15 points, NIHSS loss of consciousness 1a score ≥ 1 point E. Patients with proximal cerebral arterial occlusion (such as middle cerebral or internal carotid artery) F. Unilateral ischemic lesion of at least 2/3 of the middle cerebral artery (MCA) territory involving basal ganglia confirmed by computed tomography (CT) or magnetic resonance imaging (MRI)
* Decided to perform decompressive hemicraniectomy within 48 hours after symptom onset - Onset time was defined as the time when patients were lastly seen normal

Exclusion Criteria:

A. Premorbid modified Rankin Scale (mRS) score ≥ 2 B. Presence of other type of brain lesions including traumatic brain injury, contralateral or infratentorial infarct.

C. Absence of bilateral pupillary reflex D. Known bleeding disorder or coagulopathy E. Sepsis F. End stage malignant disease G. Pregnancy or during breast feeding H. Life expectancy less than 3 year

Ages: 19 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rankin Scale | 1 year after treatment
  Functional outcome at 1 year modified Rankin Scale of 0 to 4

SECONDARY OUTCOMES:
Mortality | 6 month, 1 year after treatment
  Mortality at 6 month, 1 year
Functional outcome | 6 month after treatment
  6 month modified Rankin Scale of 0 to 4

CONTACTS AND LOCATIONS:
Locations (1):
- Moon-Ku Han, Seongnam-si, Bundang/kyeonggido, South Korea